CLINICAL TRIAL: NCT00190671
Title: A Phase 1/2 Dose-Escalating Study of ALIMTA and Cyclophosphamide Administered Every 21 Days in Patients With Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of Pemetrexed and Cyclophosphamide Given Every 21 Days in Advanced Breast Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4029; H3E-MC-JMDV
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Breast Cancer
Keywords: Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Pemetrexed; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed 600 mg/m2 (Experimental)
  Interventions: Drug: pemetrexed; Drug: cyclophosphamide
- Pemetrexed 1800 mg/m2 (Experimental)
  Interventions: Drug: cyclophosphamide; Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — Pemetrexed: 600 mg/m2, intravenous (IV), every 21 days x 8 cycles
  Other Names: LY231514; Alimta
  Arms: Pemetrexed 600 mg/m2
Drug: cyclophosphamide — 600 mg/m2, intravenous (IV), every 21 days x 8 cycles
Drug: pemetrexed — 1800 mg/m2, intravenous (IV), every 21 days x 8 cycles
  Other Names: LY231514; Alimta
  Arms: Pemetrexed 1800 mg/m2

SUMMARY:
This is the phase 2 portion of a phase 1/2 trial, testing the use of pemetrexed and cyclophosphamide in combination for the treatment of advanced breast cancer. A single arm Phase 1 dose finding (establish maximum tolerated dose) study precedes the randomized phase 2 portion.

ELIGIBILITY:
Inclusion Criteria: - You must be female and at least 18 years old. - You must have been diagnosed with breast cancer. - Your pre-study lab tests are within study requirements. - You must be willing to take folic acid and vitamin B12. Exclusion Criteria: - You are pregnant or breastfeeding. - You have another illness that your doctor thinks would make you unable to participate. - You are currently taking aspirin or aspirin-like medicine and are unable to stop for a few days during each cycle of therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2005-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9am- 5pm Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- Austria (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Salzburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Vienna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Wels
- Czechia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Nová Ves pod Pleší
- Hungary (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Szeged
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Gdansk, Poland
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Iași
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Saint Petersburg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a Phase 1/2 study. Phase 1 determined the doses to use in the Phase 2 portion. In this 2-stage Simon's optimal design study, enrollment in the 600 mg/m2 arm was stopped at the end of Stage 1 because of lack of efficacy; ongoing patients were allowed to continue treatment. Secondary efficacy endpoints were evaluated for 1800 mg/m2 arm only.
Groups:
- Pemetrexed 600mg/m2: Pemetrexed: 600 mg/m2, intravenous, every 21 days x 8 cycles Cyclophosphamide: 600 mg/m2, intravenous, every 21 days x 8 cycles
- Pemetrexed 1800mg/m2: Pemetrexed: 1800 mg/m2, intravenous, every 21 days x 8 cycles Cyclophosphamide: 600 mg/m2, intravenous, every 21 days x 8 cycles
Period: Overall Study
Arm/Group | Pemetrexed 600mg/m2 | Pemetrexed 1800mg/m2
Started | 42 | 61
Completed | 15 | 19
Not Completed | 27 | 42
Not completed — Satisfactory Response | 4 | 7
Not completed — Lack of Efficacy | 19 | 24
Not completed — Death from Study Disease | 1 | 1
Not completed — Adverse Event | 3 | 2
Not completed — Clinical Relapse | 0 | 1
Not completed — Death from Study-Drug Toxicity | 0 | 2
Not completed — Death from Other Causes | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed 600mg/m2 | Pemetrexed 1800mg/m2 | Total
Number analyzed (Participants) | 42 | 61 | 103
Age Continuous [Median (Full Range); unit: years] | 59.0 [35 to 80] | 56.0 [32 to 81] | 58.0 [32 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 61 | 103.0
  Male | 0 | 0 | 0.0
Region of Enrollment [Number; unit: participants]
  Hungary | 11 | 11 | 22.0
  Czech Republic | 2 | 2 | 4.0
  Poland | 9 | 11 | 20.0
  Romania | 9 | 9 | 18.0
  Austria | 3 | 11 | 14.0
  Russian Federation | 8 | 17 | 25.0
Estrogen-Receptor Status [Number; unit: participants]
  Positive | 22 | 27 | 49.0
  Negative | 10 | 21 | 31.0
  Unknown | 7 | 4 | 11.0
  Missing | 3 | 9 | 12.0
Human Epidermal Growth Factor Receptor 2 (HER-2/NEU) Status [Number; unit: participants]
  Positive | 4 | 3 | 7.0
  Negative | 11 | 27 | 38.0
  Unknown | 9 | 8 | 17.0
  Not Done | 18 | 23 | 41.0
Pathological Diagnosis [Number; unit: participant]
  Inflammatory Breast Carcinoma | 7 | 10 | 17.0
  Adenocarcinoma of the Breast | 17 | 27 | 44.0
  Other | 18 | 24 | 42.0
Progesterone-Receptor Status [Number; unit: participants]
  Positive | 19 | 25 | 44.0
  Negative | 13 | 23 | 36.0
  Unknown | 7 | 4 | 11.0
  Missing | 3 | 9 | 12.0
Race/Ethnicity [Number; unit: participants]
  Caucasian | 42 | 61 | 103.0
World Health Organization Performance Status [Number; unit: participants]
  0 - Asymptomatic, fully active | 18 | 40 | 58.0
  1 - Symptomatic, fully ambulatory, light activity | 22 | 18 | 40.0
  2 - Symptomatic, ambulatory, no work activities | 2 | 3 | 5.0
Body Surface Area [Median (Full Range); unit: square meters] | 1.8 [1.4 to 2.1] | 1.7 [1.4 to 2.4] | 1.7 [1.4 to 2.4]
Height [Median (Full Range); unit: centimeters] | 160.0 [148 to 176] | 160.0 [143 to 180] | 160.0 [143 to 180]
Weight [Median (Full Range); unit: kilograms] | 71.5 [50 to 104] | 70.0 [45 to 120] | 70.0 [45 to 120]

OUTCOME MEASURES:

1. Primary Outcome: Best Tumor Response
Description: Tumor response was assessed using radiological imaging, which was repeated every 6 weeks prior to every other cycle. Confirmation of response was to occur no less than 4 weeks (28 days) after the first evidence of response.
Time Frame: baseline to measured progressive disease
Population: Number of randomized participants.
Measure: Number; unit: participants
Arm/Group | Pemetrexed 600mg/m2 | Pemetrexed 1800mg/m2
Number analyzed (Participants) | 42 | 61
participants
  Complete Response | 0 | 0
  Partial Response | 8 | 20
  Stable Disease | 18 | 26
  Progressive Disease | 13 | 8
  Unknown | 3 | 5
  Not Assessed | 0 | 2

2. Secondary Outcome: Time to Progressive Disease
Description: Time to progressive disease was defined as the time from the date of the first treatment dose to the first date of progressive disease or death from study disease.
Time Frame: baseline to measured progressive disease
Population: All randomized participants in the Phase 2 portion of the trial (enrollment in 600mg/m2 arm stopped during Phase 1 and was not continued in Phase 2). Time to disease progression was censored for 26 (42.6%) participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed 1800mg/m2
Number analyzed (Participants) | 61
months | 6.56 [5.21 to 10.92]

3. Secondary Outcome: Progression Free Survival
Description: Defined as date of first treatment dose to first date of progressive disease or death from any cause. For patients not known to have died as of data cutoff date and who did not have progressive disease, the progression free survival date was censored at last contact date.
Time Frame: baseline to measured progressive disease
Population: All randomized participants in the Phase 2 portion of the trial (enrollment in 600mg/m2 arm stopped during Phase 1 and was not continued in Phase 2). The Progression Free Survival date was censored for 22 (35.07%) participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed 1800mg/m2
Number analyzed (Participants) | 61
months | 6.26 [4.56 to 10.46]

4. Secondary Outcome: Pharmacokinetics - Maximum Observed Drug Concentration (Cmax)
Time Frame: cycle 1 (Day 1: <1 min prior to end of pemetrexed infusion; 1/2, 1, 1.5, 2, 3, 4, 6, 8, 24, 48, 72 hours after start of pemetrexed infusion)
Population: Number of participants included in the pharmacokinetic analyses.
Measure: Geometric Mean (Full Range); unit: micrograms per milliliters
Arm/Group | Pemetrexed 600mg/m2 | Pemetrexed 1800mg/m2
Number analyzed (Participants) | 5 | 9
micrograms per milliliters | 125 (15) [112 to 158] | 369 (14) [301 to 494]

5. Secondary Outcome: Pharmacokinetics - Area Under the Curve (AUC)
Description: Area under the gemcitabine concentration-time curve from zero to last quantifiable concentration [AUC(0-t)] was calculated by combination of linear and logarithmic trapezoidal methods. Linear trapezoidal method was employed up to tmax (time to reach maximal concentration), and then log trapezoidal method was used for those data after tmax.
Time Frame: as for outcome 4
Population: Number of participants included in the pharmacokinetic analyses.
Measure: Geometric Mean (Full Range); unit: hour times microgram per milliliter
Arm/Group | Pemetrexed 600mg/m2 | Pemetrexed 1800mg/m2
Number analyzed (Participants) | 5 | 9
hour times microgram per milliliter | 375 (13) [301 to 417] | 1050 (17) [877 to 1560]

6. Secondary Outcome: Pharmacokinetics - Clearance (CL)
Description: Total body clearance of drug calculated after intravenous administration.
Time Frame: as for outcome 4
Population: Number of participants included in the pharmacokinetic analyses.
Measure: Geometric Mean (Full Range); unit: milliliters per minute
Arm/Group | Pemetrexed 600mg/m2 | Pemetrexed 1800mg/m2
Number analyzed (Participants) | 5 | 9
milliliters per minute | 45.9 (15) [35.9 to 52.5] | 51.8 (27) [29 to 74.3]

7. Secondary Outcome: Pharmacokinetics - Volume of Distribution
Description: Central volume (V1) and peripheral volume (V2) of distribution.
Time Frame: as for outcome 4
Population: Number of participants included in the pharmacokinetic analyses.
Measure: Geometric Mean (Full Range); unit: Liters
Arm/Group | Pemetrexed 600mg/m2 | Pemetrexed 1800mg/m2
Number analyzed (Participants) | 5 | 9
Liters
  Central Volume of Distribution (V1) | 7.46 (16) [5.87 to 9.05] | 8.14 (25) [5.05 to 11.4]
  Peripheral Volume of Distribution (V2) | 3.58 (37) [1.95 to 4.79] | 3.33 (16) [2.51 to 4.37]

8. Secondary Outcome: Pharmacokinetics - Half-Life (t½)
Description: The half-life associated with the terminal elimination rate constant.
Time Frame: as for outcome 4
Population: Number of participants included in the pharmacokinetic analyses.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Pemetrexed 600mg/m2 | Pemetrexed 1800mg/m2
Number analyzed (Participants) | 5 | 9
hours | 4.19 [2.51 to 5.32] | 3.79 [3.09 to 4.17]

ADVERSE EVENTS:
Arm/Group | Pemetrexed 600mg/m2 | Pemetrexed 1800mg/m2
Serious Adverse Events (participants affected / at risk) | 6 | 13
Other Adverse Events (participants affected / at risk) | 38 | 59
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed 600mg/m2 | Pemetrexed 1800mg/m2
Agranulocytosis (Blood and lymphatic system disorders) | 0/42 (0) | 1/61 (1)
Anaemia (Blood and lymphatic system disorders) | 2/42 (3) | 1/61 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1/42 (1) | 0/61 (0)
Leukopenia (Blood and lymphatic system disorders) | 0/42 (0) | 2/61 (2)
Neutropenia (Blood and lymphatic system disorders) | 1/42 (2) | 2/61 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1/42 (1) | 1/61 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0/42 (0) | 1/61 (1)
Pericardial effusion (Cardiac disorders) | 1/42 (1) | 0/61 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0/42 (0) | 1/61 (1)
Melaena (Gastrointestinal disorders) | 0/42 (0) | 1/61 (1)
Fatigue (General disorders) | 1/42 (1) | 1/61 (1)
Multi-organ failure (General disorders) | 0/42 (0) | 1/61 (1)
Oedema (General disorders) | 1/42 (1) | 0/61 (0)
Hepatic failure (Hepatobiliary disorders) | 0/42 (0) | 1/61 (1)
Erysipelas (Infections and infestations) | 0/42 (0) | 1/61 (1)
Joint abscess (Infections and infestations) | 0/42 (0) | 1/61 (1)
Pneumonia (Infections and infestations) | 0/42 (0) | 1/61 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0/42 (0) | 1/61 (1)
Body temperature increased (Investigations) | 0/42 (0) | 1/61 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1/42 (1) | 1/61 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2/42 (2) | 1/61 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/42 (1) | 0/61 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed 600mg/m2 | Pemetrexed 1800mg/m2
Anaemia (Blood and lymphatic system disorders) | 3/42 (3) | 10/61 (13)
Leukopenia (Blood and lymphatic system disorders) | 8/42 (24) | 19/61 (36)
Lymphopenia (Blood and lymphatic system disorders) | 6/42 (6) | 4/61 (4)
Neutropenia (Blood and lymphatic system disorders) | 11/42 (27) | 21/61 (51)
Thrombocytopenia (Blood and lymphatic system disorders) | 3/42 (4) | 6/61 (9)
Conjunctivitis (Eye disorders) | 2/42 (3) | 7/61 (9)
Abdominal pain (Gastrointestinal disorders) | 4/42 (5) | 7/61 (7)
Abdominal pain upper (Gastrointestinal disorders) | 3/42 (3) | 2/61 (2)
Constipation (Gastrointestinal disorders) | 4/42 (4) | 3/61 (3)
Diarrhoea (Gastrointestinal disorders) | 7/42 (10) | 8/61 (9)
Nausea (Gastrointestinal disorders) | 21/42 (57) | 31/61 (79)
Stomatitis (Gastrointestinal disorders) | 1/42 (1) | 15/61 (33)
Vomiting (Gastrointestinal disorders) | 13/42 (34) | 21/61 (44)
Adverse drug reaction (General disorders) | 0/42 (0) | 4/61 (5)
Asthenia (General disorders) | 9/42 (10) | 7/61 (9)
Fatigue (General disorders) | 11/42 (25) | 20/61 (44)
Mucosal inflammation (General disorders) | 2/42 (2) | 6/61 (9)
Oedema peripheral (General disorders) | 3/42 (4) | 3/61 (4)
Pyrexia (General disorders) | 5/42 (5) | 5/61 (6)
Hypersensitivity (Immune system disorders) | 3/42 (3) | 0/61 (0)
Nasopharyngitis (Infections and infestations) | 3/42 (3) | 3/61 (3)
Alanine aminotransferase increased (Investigations) | 7/42 (9) | 13/61 (20)
Aspartate aminotransferase increased (Investigations) | 6/42 (7) | 15/61 (19)
Blood alkaline phosphatase increased (Investigations) | 9/42 (10) | 2/61 (2)
Blood lactate dehydrogenase increased (Investigations) | 3/42 (3) | 3/61 (3)
Gamma-glutamyltransferase increased (Investigations) | 3/42 (3) | 2/61 (2)
Haemoglobin decreased (Investigations) | 6/42 (11) | 6/61 (11)
Neutrophil count decreased (Investigations) | 4/42 (12) | 6/61 (16)
Platelet count decreased (Investigations) | 3/42 (3) | 4/61 (5)
White blood cell count decreased (Investigations) | 4/42 (11) | 2/61 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 0/42 (0) | 7/61 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 0/42 (0) | 7/61 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 4/42 (4) | 7/61 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 0/42 (0) | 6/61 (8)
Rash (Skin and subcutaneous tissue disorders) | 3/42 (4) | 15/61 (19)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0/42 (0) | 4/61 (4)
Hypertension (Vascular disorders) | 3/42 (4) | 3/61 (4)

LIMITATIONS AND CAVEATS:
600 mg/m2 arm discontinued at end of Phase 1 because of lack of efficacy. Enrollment in 1800 mg/m2 arm continued to Phase 2. (Phase 1 outcomes were tumor response and pharmacokinetics). Secondary efficacy endpoints analyzed for 1800 mg/m2 arm only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days